CLINICAL TRIAL: NCT05413941
Title: Internet-based Cognitive Behavioral Therapy for Black and Latino Patients With Inflammatory Bowel Disease
Brief Title: Internet-based Cognitive Behavioral Therapy in Inflammatory Bowel Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants were enrolled into this study. Study Start Date previously entered was for Aim 1 of the protocol and unrelated to this registration (see 'Detailed Description'). Primary Completion and Study Completion Dates reflect IRB closeout date.
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-14155; K12TR004411 (NIH)
Record Dates: First submitted 2022-06-07; First posted 2022-06-10 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Bowel Diseases; Psychological Distress
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internet-based Cognitive Behavioral Therapy (Experimental)
  Interventions: Behavioral: Internet-based Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Internet-based Cognitive Behavioral Therapy — Cognitive behavioral therapy (CBT) is a form of psychotherapy in which individuals are taught to identify and modify maladaptive thinking and behavior to improve their psychological status and coping skills. CBT in this trial will be delivered digitally (internet-based).

SUMMARY:
While people of color are an increasing segment of the inflammatory bowel disease (IBD) population, they are currently underrepresented in research, including studies of psychological distress. Appreciation for psychological distress (anxiety, depression, perceived stress) as a driver of IBD activity has led to increased efforts to integrate psychological interventions into IBD medical care. Cognitive behavioral therapy (CBT) is the most studied psychotherapeutic approach in IBD and the one that suggests improvements in mental health and quality of life in those with elevated psychological distress. There are unanswered questions in the use of CBT in IBD: how to leverage digital technology to deliver CBT through internet-based cognitive behavioral therapy (iCBT); how do we consider the social context of individuals from racial and ethnic minority groups who may experience distinct social and structural barriers to acceptance and use of psychological interventions? Thus, this study will qualitatively analyze how factors, such as digital access, mental health stigma, and lived experience with IBD and as racial or ethnic minority influence attitudes toward mental health and iCBT in a cohort of Black and Latino IBD patients with elevated psychological distress. Results will lead to adaptation of a CBT program into an iCBT app to be tested for acceptance/use and to explore effects on psychological and disease-related factors.

DETAILED DESCRIPTION:
The clinical trial component of this study (Aim 3) was never conducted. Only Aim 1, consisting of an assessment of the factors influencing acceptance and use of iCBT via semi-structured interviews, and which did not meet the definition of a clinical trial, was conducted as part of this study. The clinical trial component associated with this study, the internet-based cognitive therapy (iCBT), is being conducted as part of the "Digital Mind Body Intervention Among Black and Hispanic Patients Living With Inflammatory Bowel Disease (DMBI)," NCT06510296 (ID: 2024-16064) clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as Black or Hispanic/Latino
* diagnosis of Crohn's disease or ulcerative colitis
* ability to provide informed consent in English
* basic computer skills (i.e. ability to self-complete online questionnaire)
* elevated psychological distress

Exclusion Criteria:

* severe psychological distress
* active suicidality, past suicide attempt, or psychiatric hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | 8 weeks
  Proportion of eligible patients who enroll into the trial
Adherence Rate | 8 weeks
  Number of activities and weekly sessions completed

SECONDARY OUTCOMES:
Illness Perception | 8 weeks
  Cognitive and emotional representations formed about one's illness measured via Brief Illness Perception Questionnaire (minimum 0, maximum 80; higher scores indicate more severe illness impact)
Self-efficacy | 8 weeks
  A task-specific construct of the perception of one's ability to manage a given situation measured via PROMIS-Self Efficacy in Managing Emotions questionnaire (T score 50 is the mean, higher scores indicate greater self efficacy)
Coping | 8 weeks
  Manner of dealing with stress measured via Brief Resilient Coping Scale (minimum 4, maximum 20; higher scores indicate greater resilience)
Crohn's Activity | 8 weeks
  Level of symptomatic disease measured via Short Crohn's Disease Activity index
Ulcerative Colitis Activity | 8 weeks
  Level of symptomatic disease measured via Simple Clinical Colitis Activity index
Interleukin-6 level | 8 weeks
  Inflammatory biomarker
Health related quality of life | 8 weeks
  Quality of life measured via PROMIS-29 questionnaire (mean T score is 50, higher scores indicate higher degree of measured trait)

CONTACTS AND LOCATIONS:
Overall Officials: Ruby Greywoode, MD, Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: No